CLINICAL TRIAL: NCT01477684
Title: Documentation of In-flight Medical Emergencies With Medical Incident Report Forms.
Status: Completed | Type: Observational
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Michael Sand, Principal Investigator, Ruhr University of Bochum
Other Study IDs: FM1
Record Dates: First submitted 2011-11-18; First posted 2011-11-22 (Estimated); Last update posted 2012-10-16 (Estimated); Status verified 2012-10

CONDITIONS: In-flight Medical Emergency

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to perform a descriptive, content-based analysis on the different forms of documentation for in-flight medical emergencies that are currently provided in the emergency medical kits on board commercial airlines.

ELIGIBILITY:
Inclusion Criteria:

* medical incident report form

Exclusion Criteria:

* no medical incident report form

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: medical incident report forms
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2011-10; Primary Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dermatology, Venereology and Allergology, Ruhr-University Bochum, Bochum, North Rhine-Westphalia, Germany

REFERENCES:
- [Result] Sand M, Morrosch S, Sand D, Altmeyer P, Bechara FG. Medical emergencies on board commercial airlines: is documentation as expected? Crit Care. 2012 Dec 12;16(2):R42. doi: 10.1186/cc11238. PMID 22397530